CLINICAL TRIAL: NCT04421417
Title: Early-term Effects of Microfracture on Tendon Vascularity and Healing in Arthroscopic Treatment of Chronic Rotator Cuff Tears: A Prospective Randomized Trial
Brief Title: The Effect of Microfracture Procedure on Rotator Cuff Tendon Healing
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped due to COVID-19 related issues. Collected data could be present as pilot trial.
Sponsor: Göker Utku değer (Other)
Responsible Party: Sponsor-Investigator, Göker Utku değer, Research assistant, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-78167
Record Dates: First submitted 2020-06-02; First posted 2020-06-09 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Rotator Cuff Tears; Micro Fracture
Keywords: Superb microvascular imaging; Rotator Cuff Tears; Micro Fracture
MeSH Terms: conditions — Rotator Cuff Injuries; Fractures, Stress

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Arthroscopic Rotator Cuff Repair (Active Comparator)
  Interventions: Procedure: Standard Arthroscopic Rotator Cuff Repair
- Microfracture and Arthroscopic Rotator Cuff Repair (Experimental)
  Interventions: Procedure: Microfracture + Standard Arthroscopic Rotator Cuff Repair

INTERVENTIONS:
Procedure: Microfracture + Standard Arthroscopic Rotator Cuff Repair — drilling of rotator cuff footprint area on humerus and standard arthroscopic rotator cuff repair
  Arms: Microfracture and Arthroscopic Rotator Cuff Repair
Procedure: Standard Arthroscopic Rotator Cuff Repair — Standard Arthroscopic Rotator Cuff Repair
  Arms: Standard Arthroscopic Rotator Cuff Repair

SUMMARY:
Patients with complaints of shoulder pain or limitation of motion and had rotator cuff rupture diagnosed with magnetic resonance imaging will be analyzed and the patients with surgical indication will be included in a randomized fashion. One group of patient will undergo standard arthroscopic rotator cuff repair, while the other group will have microfracture procedure in addition to the standard arthroscopic repair. Before the operation, functional and clinical conditions will be recorded with Constant and American Shoulder and Elbow Surgeons Shoulder Score (ASES) universal shoulder scoring systems and Visual Analogue Scale(VAS) pain scale. The blood supply and healing of the tendon in the repair area will be compared by the doppler ultrasound (superb microvascular imaging) at the 2nd, 4th, 8th and 12th week after the operation. Post-operative clinical, functional status and pain levels will be evaluated with Constant, ASES and VAS pain scales at 24th week.

ELIGIBILITY:
Inclusion Criteria:

* degenerative rotator cuff tears

Exclusion Criteria:

* traumatic rotator cuff tears
* rheumatoid diseases
* previous surgery of rotator cuff tendon
* glenohumeral arthritis
* acromioclavicular arthritis

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
assessing early change of tendon and footprint area vascularity | 4th week
  we will evaluate it by superb microvascular imaging via ultrasound, this ultrasound software give us quantitative value of vascularity
assessing early change of tendon and footprint area vascularity | 8th week
  we will evaluate it by superb microvascular imaging via ultrasound, this ultrasound software give us quantitative value of vascularity
assessing early change of tendon and footprint area vascularity | 12th week
  we will evaluate it by superb microvascular imaging via ultrasound, this ultrasound software give us quantitative value of vascularity

SECONDARY OUTCOMES:
functional outcome | 24th week
  This entity will be asses by functional scoring systems.These are American Shoulder and Elbow Surgeons Shoulder Score (ASES) and Constant Shoulder Score. The ASES is a composite instrument, requiring both a physician assessment and a patient-completed portion; however, it is commonly presented as solely the patient-reported survey. This includes a section on pain (7 items) and a section on activities of daily living (10 items). Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition. Constant Score was designed to assess the functional state of a normal, a diseased, or a treated shoulder.The Constant score contains both physician-completed and patient-reported portions. The four domains include pain (15 possible points), activities of daily living (20 possible points), mobility (40 possible points), and strength (25 possible points). Scores range from 0 points (most disability) to 100 points (least disability).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University- Cerrahpasa Cerrahpasa Medical Faculty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodeo SA, Delos D, Williams RJ, Adler RS, Pearle A, Warren RF. The effect of platelet-rich fibrin matrix on rotator cuff tendon healing: a prospective, randomized clinical study. Am J Sports Med. 2012 Jun;40(6):1234-41. doi: 10.1177/0363546512442924. Epub 2012 Apr 10. PMID 22495146
- [Background] Zumstein MA, Rumian A, Lesbats V, Schaer M, Boileau P. Increased vascularization during early healing after biologic augmentation in repair of chronic rotator cuff tears using autologous leukocyte- and platelet-rich fibrin (L-PRF): a prospective randomized controlled pilot trial. J Shoulder Elbow Surg. 2014 Jan;23(1):3-12. doi: 10.1016/j.jse.2013.08.017. PMID 24331121
- [Background] Milano G, Saccomanno MF, Careri S, Taccardo G, De Vitis R, Fabbriciani C. Efficacy of marrow-stimulating technique in arthroscopic rotator cuff repair: a prospective randomized study. Arthroscopy. 2013 May;29(5):802-10. doi: 10.1016/j.arthro.2013.01.019. Epub 2013 Mar 21. PMID 23522987
- [Background] Osti L, Del Buono A, Maffulli N. Microfractures at the rotator cuff footprint: a randomised controlled study. Int Orthop. 2013 Nov;37(11):2165-71. doi: 10.1007/s00264-013-1952-z. Epub 2013 Jun 13. PMID 23760681
- [Background] Bilsel K, Yildiz F, Kapicioglu M, Uzer G, Elmadag M, Pulatkan A, Esrefoglu M, Bozdag E, Milano G. Efficacy of bone marrow-stimulating technique in rotator cuff repair. J Shoulder Elbow Surg. 2017 Aug;26(8):1360-1366. doi: 10.1016/j.jse.2017.02.014. Epub 2017 Apr 7. PMID 28395947